CLINICAL TRIAL: NCT02966834
Title: A Randomized, Double-blind, Multi-dose, Placebo-controlled Study to Evaluate the Efficacy, Safety and Tolerability of GSK2330672 Administration for the Treatment of Pruritus in Patients With Primary Biliary Cholangitis (GLIMMER: GSK2330672 triaL of IBAT Inhibition With Multidose Measurement for Evaluation of Response)
Brief Title: Dose Response Study of GSK2330672 for the Treatment of Pruritus in Participants With Primary Biliary Cholangitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 201000; 2016-002416-41 (EudraCT Number)
Record Dates: First submitted 2016-11-15; First posted 2016-11-17 (Estimated); Results first posted 2021-05-04 (Actual); Last update posted 2021-05-04 (Actual); Status verified 2021-04

CONDITIONS: Cholestasis
Keywords: linerixibat; PBC; itch; GSK2330672; GLIMMER; primary biliary cholangitis; pruritus
MeSH Terms: conditions — Cholestasis; Pruritus; Liver Cirrhosis, Biliary | interventions — 3-((((3R,5R)-3-butyl-3-ethyl-7-(methyloxy)-1,1-dioxido-5-phenyl-2,3,4,5-tetrahydro-1,4-benzothiazepin-8-yl)methyl)amino)pentanedioic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Placebo (Placebo Comparator): Participants will receive matching placebo
  Interventions: Drug: Placebo
- GSK2330672 20 mg once daily (Experimental): Participants will receive GSK2330672 and matching placebo to maintain blind
  Interventions: Drug: Placebo; Drug: GSK2330672
- GSK2330672 90 mg once daily (Experimental): Participants will receive GSK2330672 and matching placebo to maintain blind
  Interventions: Drug: Placebo; Drug: GSK2330672
- GSK2330672 180 mg once daily (Experimental): Participants will receive GSK2330672 and matching placebo to maintain blind
  Interventions: Drug: Placebo; Drug: GSK2330672
- GSK2330672 40 mg twice daily (Experimental): Participants will receive GSK2330672 and matching placebo to maintain blind
  Interventions: Drug: Placebo; Drug: GSK2330672
- GSK2330672 90 mg twice daily (Experimental): Participants will receive GSK2330672 and matching placebo to maintain blind
  Interventions: Drug: Placebo; Drug: GSK2330672

INTERVENTIONS:
Drug: Placebo — GSK2330672 matching placebo will be supplied as white film-coated tablets.
Drug: GSK2330672 — GSK2330672 will be supplied in 2 dose strengths of 10 mg and 45 mg white film-coated tablets.
  Arms: GSK2330672 180 mg once daily; GSK2330672 20 mg once daily; GSK2330672 40 mg twice daily; GSK2330672 90 mg once daily; GSK2330672 90 mg twice daily

SUMMARY:
This study is being conducted to evaluate the efficacy, safety and tolerability of GSK2330672 administration for the treatment of pruritus (itch) in participants with primary biliary cholangitis (PBC). Participants will receive either placebo or one of the 4 dose regimens of GSK2330672 (20 milligram [mg], 90 mg or 180 mg taken once daily or 90 mg twice daily). Participants on GSK2330672 will also receive placebo tablets to maintain blinding. The study has a prospectively defined adaptive design that will utilize interim data to further inform and potentially optimize the doses under investigation. Hence, additional dose regimen may be added during study. The total duration of a participant in the study will be up to 45 days of screening and 24 weeks of study including follow-up.

ELIGIBILITY:
Inclusion Criteria

* Participant must be 18 to 80 years of age inclusive, at the time of signing the informed consent.
* Participants who have proven PBC, as demonstrated by having at least 2 of the following: History of sustained increased ALP levels >ULN first recognized at least 6 months prior to the Screening Visit (Sustained ALP elevations at the time of Screening is not required, recognizing that the ALP may have decreased after institution of ursodeoxycholic acid (UDCA) therapy as described in inclusion number 4). Documented positive anti-mitochondrial antibody (AMA) titer (>1:40 titer on immunofluorescence or M2 positive by enzyme-linked immunosorbent assay) or PBC-specific antinuclear antibodies (antinuclear dot and/or nuclear rim positive). Liver biopsy (at any time in the past) consistent with PBC.
* Participants must rate their itch severity as being >=4 on a 0 to 10 point scale for the majority of time (at least half the days, as recalled by the participant) during the 8 weeks prior to the Screening Visit. Periods of low itch or no itch are acceptable as long as the worst daily itch score is >=4 on the majority of days.
* Participants who are currently taking UDCA should be on stable doses of UDCA for >8 weeks at time of screening. Participants not taking UDCA due to intolerance may be enrolled 8 weeks after their last dose of UDCA. No changes or discontinuation is permitted until completion of the Main Study Period.
* Male and/or female: Female participants- A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies: Not a woman of childbearing potential (WOCBP) or a WOCBP who agrees to follow the contraceptive guidance during the treatment period and until at least 4 weeks after the last dose of study treatment.
* Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.

Exclusion Criteria

* Screening total bilirubin >2x ULN. Total bilirubin >2x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35 percent (%).
* Screening ALT or AST >6x ULN.
* Screening eGFR <45 milliliter (mL)/minute/1.73 square meter (m^2) based on the CKD-EPI.
* History or presence of hepatic decompensation (e.g., variceal bleeds, encephalopathy or ascites).
* Presence of actively replicating viral hepatitis due to hepatitis B or C virus (HBV, HCV) infection, and/or confirmed hepatocellular carcinoma or biliary cancer. Other hepatic conditions ( e.g., primary sclerosing cholangitis [PSC], alcoholic liver disease, autoimmune hepatitis, non-alcoholic steatohepatitis [NASH] ) are permitted if PBC is the dominant liver injury in the investigator's opinion.
* Current diarrhea.
* Current symptomatic cholelithiasis or inflammatory gall bladder disease. Participants with history of cholecystectomy >=3 months before screening may be eligible for enrolment.
* Any current medical condition (e.g. psychiatric disorder, senility or dementia), which may affect the participant's ability to comply with the protocol specified procedures.
* Initiation or increase in dose of colchicine, methotrexate, azathioprine, or systemic corticosteroids in the 2 months prior to screening. If a change in dose in any of these medications is anticipated during the course of the study, the participant should be excluded.
* Initiation or increase in dose of bezafibrate or fenofibrate at any time during the 3 months prior to screening. Participants may join the study on stable doses of these medications, but no change or discontinuation is permitted until completion of the Main Study Period.
* Initiation or increase in dose of any of the following in the 8 weeks prior to screening: rifampicin, naltrexone, naloxone, nalfurafine, or sertraline. Participants may join the study on stable or decreased doses of these medications, but no change in dose is permitted until completion of the Main Study Period.
* Bile acid binding resin use: a participant must discontinue use of cholestyramine, colesevelam, colestipol or colestimide prior to the start of the Initial Study Period (no later than Day-2). Note: these drugs may be administered after completion of the Main Study Period, if clinically indicated.
* Obeticholic acid use: a participant must discontinue use of obeticholic acid at least 8 weeks prior to the start of the Initial Study Period and may not restart until after the end of the study.
* Administration of any other Inhibitor of the Human Ileal Bile Acid Transporter (IBAT) in the 3 months prior to screening.
* Current enrolment or participation within the 8 weeks before start of the Initial Study Period, in any other clinical study involving an investigational study treatment.
* QT interval corrected for heart rate QTc >480 millisecond (msec).
* History of sensitivity to the study treatment or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GlaxoSmithKline (GSK) Medical Monitor, contraindicates their participation in the study.
* History of regular alcohol consumption within 6 months of the study defined as an average weekly intake of >21 units for males or >14 units for females. One unit is equivalent to 8 gram of alcohol: a half-pint (approximately 240 mL) of beer, 1 glass (125 mL) of wine or 1 measure (25 mL) of spirits.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2017-01-11 (Actual); Primary Completion 2020-04-15 (Actual); Study Completion 2020-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (62):
- United States (9):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Novi, Michigan
  - GSK Investigational Site, Manhasset, New Jersey
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Allentown, Pennsylvania
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Seattle, Washington
- Australia (4):
  - GSK Investigational Site, Camperdown, New South Wales
  - GSK Investigational Site, Herston, Queensland
  - GSK Investigational Site, Prahran, Victoria
  - GSK Investigational Site, Nedlands, Western Australia
- Canada (6):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (5):
  - GSK Investigational Site, Clermont-Ferrand
  - GSK Investigational Site, Grenoble
  - GSK Investigational Site, Lille
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Pessac
- Germany (3):
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Homburg, Saarland
  - GSK Investigational Site, Hamburg
- Italy (5):
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Monza (MB), Lombardy
  - GSK Investigational Site, Florence, Tuscany
  - GSK Investigational Site, Padua, Veneto
- Japan (10):
  - GSK Investigational Site, Chiba
  - GSK Investigational Site, Fukui
  - GSK Investigational Site, Gunma
  - GSK Investigational Site, Hiroshima
  - GSK Investigational Site, Hokkaido
  - GSK Investigational Site, Kagawa
  - GSK Investigational Site, Kanagawa
  - GSK Investigational Site, Nagasaki
  - GSK Investigational Site, Osaka
  - GSK Investigational Site, Tokyo
- Poland (5):
  - GSK Investigational Site, Częstochowa
  - GSK Investigational Site, Katowice
  - GSK Investigational Site, Mysłowice
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Spain (4):
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
- United Kingdom (11):
  - GSK Investigational Site, Basingstoke
  - GSK Investigational Site, Edgbaston
  - GSK Investigational Site, Glasgow
  - GSK Investigational Site, Liverpool
  - GSK Investigational Site, London
  - GSK Investigational Site, Manchester
  - GSK Investigational Site, Middlesbrough
  - GSK Investigational Site, Newcastle upon Tyne
  - GSK Investigational Site, Nottingham
  - GSK Investigational Site, Plymouth
  - GSK Investigational Site, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study will be made available via the Clinical Study Data Request site.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD will be made available within 6 months of publishing the results of the primary endpoints, key secondary endpoints and safety data of the study.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: http://clinicalstudydatarequest.com

REFERENCES:
- [Derived] Carreno F, Karatza E, Mehta R, Collins J, Austin D, Swift B. Population Dose-Response-Time Analysis of Itch Reduction and Patient-Reported Tolerability Supports Phase III Dose Selection for Linerixibat. Clin Pharmacol Ther. 2024 Feb;115(2):288-298. doi: 10.1002/cpt.3103. Epub 2023 Dec 3. PMID 37953500
- [Derived] Tanaka A, Atsukawa M, Tsuji K, Notsumata K, Suyama A, Ito H, Das S, von Maltzahn R, McLaughlin MM. Japanese subgroup analysis of GLIMMER: A global Phase IIb study of linerixibat for the treatment of cholestatic pruritus in patients with primary biliary cholangitis. Hepatol Res. 2023 Jul;53(7):629-640. doi: 10.1111/hepr.13895. Epub 2023 Mar 13. PMID 36852705
- [Derived] Levy C, Kendrick S, Bowlus CL, Tanaka A, Jones D, Kremer AE, Mayo MJ, Haque N, von Maltzahn R, Allinder M, Swift B, McLaughlin MM, Hirschfield GM; GLIMMER Study Group. GLIMMER: A Randomized Phase 2b Dose-Ranging Trial of Linerixibat in Primary Biliary Cholangitis Patients With Pruritus. Clin Gastroenterol Hepatol. 2023 Jul;21(7):1902-1912.e13. doi: 10.1016/j.cgh.2022.10.032. Epub 2022 Nov 4. PMID 36343847

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted across 66 centers in 10 countries. The 40 milligrams (mg) twice daily dose group was added and recruitment into the 20 mg twice daily dose group was discontinued following the pre-specified interim analysis.
Pre-assignment Details: A total of 147 adult participants were randomized in this study.
Groups:
- Placebo: Eligible participants were randomized to receive GSK2330672 matching placebo via oral route for 16 weeks including the Main Study Period and Final Study period. Participants were then followed up for 4 weeks.
- GSK2330672 20 mg QD: Eligible participants were randomized to receive GSK2330672 20 milligrams (mg) once daily (QD) for 12 weeks in the Main Study period followed by matching placebo for 4 weeks in the Final Study period. Participants were then followed up for 4 weeks. All doses were administered via oral route.
- GSK2330672 90 mg QD: Eligible participants were randomized to receive GSK2330672 90 mg QD for 12 weeks in the Main study period followed by matching placebo for 4 weeks in the Final Study Period. Participants were then followed up for 4 weeks. All doses were administered via oral route.
- GSK2330672 180 mg QD: Eligible participants were randomized to receive GSK2330672 180 mg QD for 12 weeks in the Main study period followed by matching placebo for 4 weeks in the Final study period. Participants were then followed up for 4 weeks. All doses were administered via oral route.
- GSK2330672 40 mg BID: Eligible participants were randomized to receive GSK2330672 40 mg twice daily (BID) for 12 weeks in the Main study period followed by matching placebo for 4 weeks in the Final study period. Participants were then followed up for 4 weeks. All doses were administered via oral route.
- GSK2330672 90 mg BID: Eligible participants were randomized to receive GSK2330672 90 mg BID for 12 weeks in the Main study period followed by matching placebo for 4 weeks in the Final Study Period. Participants were then followed up for 4 weeks All doses were administered via oral route.
Period: Main Study Period (Up to 12 Weeks)
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Started | 36 | 16 | 23 | 27 | 23 | 22
Completed | 35 | 16 | 19 | 19 | 22 | 17
Not Completed | 1 | 0 | 4 | 8 | 1 | 5
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Discontinued study treatment and entered follow-up | 0 | 0 | 4 | 8 | 0 | 5
Period: Final Study Period (Up to 4 Weeks)
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Started | 35 | 16 | 19 | 19 | 21 (One participant did not enter Final Study Period.) | 17
Completed | 35 | 16 | 19 | 19 | 21 | 17
Not Completed | 0 | 0 | 0 | 0 | 0 | 0
Period: Follow-up (Up to 4 Weeks)
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Started | 35 | 16 | 23 (4 participants discontinued study treatment in Main study period and directly entered follow-up.) | 27 (8 participants discontinued study treatment in Main Study period and directly entered follow-up.) | 22 (1 participant who completed main study period directly entered follow-up in this arm) | 22 (5 participants discontinued study treatment in Main study period and directly entered follow-up)
Completed | 35 | 16 | 22 | 22 | 22 | 21
Not Completed | 0 | 0 | 1 | 5 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics is presented for Safety Population which consisted of all randomized participants who took at least one dose of randomized study treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID | Total
Number analyzed (Participants) | 36 | 16 | 23 | 27 | 23 | 22 | 147
Age, Continuous [Mean (Standard Deviation); unit: Years] | 54.4 (11.06) | 58.5 (7.35) | 52.5 (12.32) | 58.9 (11.10) | 55.6 (11.23) | 56.2 (11.32) | 55.8 (11.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 16 | 21 | 25 | 22 | 20 | 138
  Male | 2 | 0 | 2 | 2 | 1 | 2 | 9
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaskan Native | 0 | 0 | 0 | 0 | 1 | 0 | 1
  Asian - Japanese Heritage | 8 | 6 | 6 | 7 | 4 | 7 | 38
  White - White/Caucasian/European Heritage | 26 | 10 | 17 | 19 | 16 | 15 | 103
  Multiple | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Unknown | 2 | 0 | 0 | 0 | 2 | 0 | 4

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline at Week 16 in the Mean Worst Daily Itch Score
Description: Participants were required to score the severity of their itching using a 0-10 numerical rating scale (NRS) where 0 represents no itching and 10 indicates the worst imaginable itching. The Worst Daily Itch Score is the most severe (highest) NRS recorded on a given day. Mean Worst Daily Itch score was calculated as the average of the worst daily itch scores provided in the 7 days prior to the Week 16 visit. Baseline is the average of the scores in the 7 days prior to the Week 4 (Visit 3 [V3]). Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Analysis was done using Analysis of covariance (ANCOVA) including treatment group and centered Mean Worst Daily Itch score at Baseline.
Time Frame: Baseline and Week 16
Population: Intent-to-Treat (ITT) Population comprised of all randomized participants who received at least one dose of study treatment, had a Baseline and at least one on-treatment assessment. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 35 | 16 | 20 | 22 | 22 | 21
Scores on a scale | -1.73 [-2.44 to -1.01] | -2.19 [-3.26 to -1.12] | -2.60 [-3.55 to -1.65] | -2.60 [-3.51 to -1.70] | -2.86 [-3.76 to -1.95] | -2.25 [-3.19 to -1.32]
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = -0.47, 95% CI 2-sided [-1.75 to 0.82]
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = -0.88, 95% CI 2-sided [-2.07 to 0.31]
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = -0.88, 95% CI 2-sided [-2.03 to 0.28]
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = -1.13, 95% CI 2-sided [-2.29 to 0.03]
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = -0.53, 95% CI 2-sided [-1.71 to 0.65]

2. Secondary Outcome: Mean Change From Baseline at Week 16 in Primary Biliary Cholangitis-40 (PBC-40) Scale
Description: PBC-40 is a disease-specific health-related quality of life (HRQoL) questionnaire for use in PBC participants. It consists of 40 questions arranged in 6 domains with 3 to 11 questions in each domain. Each question is scored from 1 (least impact) to 5 (greatest impact). All questions within a domain are summed to obtain individual domain score. Domains were: Symptoms (7 questions) with score range 7-35, Itch (3 questions) with score range 3-15, Fatigue (11 questions) with score range 11-55, Cognitive (6 questions) with score range 6-30, Emotional (3 questions) with score range 3-15, and Social (10 questions) with score range 10-50. Higher scores for individual domains represent a poor quality of life. Baseline is the assessment performed at Week 4 (V3) which is conducted prior to first dosing of randomized medication that evening. Change from Baseline was calculated as post-Baseline value minus Baseline value. Analysis was performed using ANCOVA including treatment group and Baseline.
Time Frame: Baseline and at Week 16
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 35 | 16 | 21 | 22 | 22 | 20
Scores on a scale
  Symptoms | 0.2 [-1.0 to 1.4] | 0.4 [-1.3 to 2.2] | 0.7 [-0.8 to 2.3] | -0.9 [-2.4 to 0.6] | 0.3 [-1.2 to 1.8] | 0.2 [-1.4 to 1.8]
  Itch | -2.3 [-3.3 to -1.4] | -1.9 [-3.3 to -0.4] | -2.6 [-3.9 to -1.3] | -2.7 [-3.9 to -1.4] | -3.4 [-4.6 to -2.1] | -2.7 [-4.0 to -1.4]
  Fatigue | -1.8 [-4.0 to 0.4] | -2.4 [-5.6 to 0.7] | -1.1 [-3.8 to 1.7] | 1.7 [-1.0 to 4.5] | -0.1 [-2.8 to 2.6] | -1.8 [-4.6 to 1.1]
  Cognitive | -0.3 [-1.7 to 1.1] | -0.3 [-2.4 to 1.8] | -0.9 [-2.7 to 0.9] | -0.1 [-1.9 to 1.6] | 0.1 [-1.6 to 1.9] | -0.1 [-2.0 to 1.7]
  Emotional | -0.5 [-1.2 to 0.1] | -1.4 [-2.4 to -0.4] | -0.4 [-1.3 to 0.5] | -0.6 [-1.5 to 0.3] | -1.4 [-2.2 to -0.5] | -0.6 [-1.5 to 0.3]
  Social | -0.8 [-2.3 to 0.8] | -0.5 [-2.7 to 1.8] | 0.4 [-1.5 to 2.4] | -0.6 [-2.5 to 1.3] | -3.1 [-5.1 to -1.2] | -1.0 [-3.0 to 1.0]
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = 0.2, 95% CI 2-sided [-1.9 to 2.3] — Symptoms
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = 0.5, 95% CI 2-sided [-1.5 to 2.5] — Symptoms
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = -1.1, 95% CI 2-sided [-3.1 to 0.8] — Symptoms
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = 0.1, 95% CI 2-sided [-1.8 to 2.0] — Symptoms
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = 0.0, 95% CI 2-sided [-2.0 to 1.9] — Symptoms
Statistical Analysis 6: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = 0.5, 95% CI 2-sided [-1.3 to 2.2] — Itch
Statistical Analysis 7: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = -0.3, 95% CI 2-sided [-1.8 to 1.3] — Itch
Statistical Analysis 8: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = -0.3, 95% CI 2-sided [-1.9 to 1.2] — Itch
Statistical Analysis 9: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = -1.0, 95% CI 2-sided [-2.6 to 0.5] — Itch
Statistical Analysis 10: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = -0.3, 95% CI 2-sided [-1.9 to 1.3] — Itch
Statistical Analysis 11: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = -0.6, 95% CI 2-sided [-4.5 to 3.2] — Fatigue
Statistical Analysis 12: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Median Difference (Net) = 0.7, 95% CI 2-sided [-2.8 to 4.2] — Fatigue
Statistical Analysis 13: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = 3.5, 95% CI 2-sided [0.0 to 7.0] — Fatigue
Statistical Analysis 14: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = 1.7, 95% CI 2-sided [-1.8 to 5.1] — Fatigue
Statistical Analysis 15: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = 0.0, 95% CI 2-sided [-3.6 to 3.6] — Fatigue
Statistical Analysis 16: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = 0.0, 95% CI 2-sided [-2.5 to 2.6] — Cognitive
Statistical Analysis 17: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = -0.6, 95% CI 2-sided [-2.9 to 1.7] — Cognitive
Statistical Analysis 18: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = 0.2, 95% CI 2-sided [-2.1 to 2.5] — Cognitive
Statistical Analysis 19: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = 0.5, 95% CI 2-sided [-1.8 to 2.8] — Cognitive
Statistical Analysis 20: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = 0.2, 95% CI 2-sided [-2.2 to 2.5] — Cognitive
Statistical Analysis 21: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = -0.9, 95% CI 2-sided [-2.1 to 0.4] — Emotional
Statistical Analysis 22: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = 0.2, 95% CI 2-sided [-0.9 to 1.3] — Emotional
Statistical Analysis 23: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = -0.1, 95% CI 2-sided [-1.2 to 1.1] — Emotional
Statistical Analysis 24: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = -0.8, 95% CI 2-sided [-1.9 to 0.3] — Emotional
Statistical Analysis 25: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = 0.0, 95% CI 2-sided [-1.2 to 1.1] — Emotional
Statistical Analysis 26: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = 0.3, 95% CI 2-sided [-2.4 to 3.0] — Social
Statistical Analysis 27: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = 1.2, 95% CI 2-sided [-1.3 to 3.7] — Social
Statistical Analysis 28: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = 0.2, 95% CI 2-sided [-2.3 to 2.7] — Social
Statistical Analysis 29: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = -2.4, 95% CI 2-sided [-4.8 to 0.1] — Social
Statistical Analysis 30: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = -0.2, 95% CI 2-sided [-2.8 to 2.4] — Social

3. Secondary Outcome: Mean Change From Baseline at Week 16 in Serum Alkaline Phosphatase (ALP) Concentrations, in Participants With High Risk of PBC Progression
Description: Criteria for high risk of PBC progression is defined as serum ALP concentrations more than or equal to (>=)1.67 times upper limit of normal (ULN) range and/or total bilirubin concentrations more than (>)ULN at Day 1. Baseline is the assessment performed at Week 4 (V3), or if missing then Visit 2 (Day 1) or Visit 1 (Screening), excluding unscheduled visits. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Analysis was performed using ANCOVA including treatment group and Baseline.
Time Frame: Baseline and at Week 16
Population: High Risk Population comprised of subset of the ITT population who were assigned to the High Risk stratum for randomization (based upon serum ALP concentrations >=1.67 times ULN and/or total bilirubin concentrations >ULN at Day 1 (Visit 2). Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: International units per Liter
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 11 | 5 | 11 | 7 | 6 | 5
International units per Liter | 49.1 [-29.3 to 127.6] | -57.7 [-179.6 to 64.3] | -38.2 [-117.0 to 40.5] | 49.6 [-49.1 to 148.2] | -29.2 [-136.7 to 78.3] | 19.1 [-97.7 to 136.0]
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = -106.8, 95% CI 2-sided [-251.7 to 38.2]
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = -87.4, 95% CI 2-sided [-198.5 to 23.8]
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = 0.4, 95% CI 2-sided [-125.6 to 126.5]
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = -78.3, 95% CI 2-sided [-211.5 to 54.8]
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = -30.0, 95% CI 2-sided [-170.7 to 110.7]

4. Secondary Outcome: Number of Participants With Serum ALP Concentrations Less Than (<)1.67 Times ULN and Total Bilirubin Concentrations Less Than or Equal to (<=) ULN at Week 16
Description: Number of participants with ALP < 1.67 times ULN and total bilirubin <= ULN at Week 16 is presented. The endpoint was analyzed in Restricted High Risk Population.
Time Frame: At Week 16
Population: Restricted High Risk Population comprised of a subset of the High Risk population, i.e. all those participants assigned to the High Risk stratum for randomization who met the ALP/bilirubin criteria at both Visit 2 (Day 1) and Visit 3 (Week 4).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 11 | 5 | 9 | 9 | 6 | 7
Participants | 0 | 0 | 0 | 0 | 0 | 1

5. Secondary Outcome: Mean Change From Baseline at Week 16 in Serum Alanine Aminotransferase (ALT) Among Those With a High Risk of PBC Progression
Description: Baseline is the assessment performed at Week 4 (V3), or if missing then Visit 2 or Visit 1, excluding unscheduled visits. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Analysis was performed using ANCOVA model including Treatment group and Baseline.
Time Frame: Baseline and at Week 16
Population: High Risk Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: International Units per Liter
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 11 | 5 | 11 | 7 | 6 | 5
International Units per Liter | 13.0 [-7.9 to 33.9] | -8.4 [-39.5 to 22.7] | 0.3 [-20.7 to 21.2] | -2.0 [-29.0 to 25.1] | -13.5 [-42.8 to 15.9] | 13.2 [-17.4 to 43.7]
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = -21.4, 95% CI 2-sided [-58.4 to 15.5]
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = -12.7, 95% CI 2-sided [-41.9 to 16.4]
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = -15.0, 95% CI 2-sided [-49.9 to 20.0]
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = -26.5, 95% CI 2-sided [-63.3 to 10.4]
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = 0.2, 95% CI 2-sided [-36.7 to 37.1]

6. Secondary Outcome: Mean Change From Baseline at Week 16 in Serum Aspartate Aminotransferase (AST) Among Those With a High Risk of PBC Progression
Description: as for outcome 5
Time Frame: Baseline and at Week 16
Population: High Risk Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: International Units per Liter
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 11 | 5 | 11 | 7 | 6 | 5
International Units per Liter | 13.96 [-4.55 to 32.46] | -6.04 [-34.20 to 22.12] | -10.75 [-28.90 to 7.40] | -8.66 [-32.24 to 14.93] | -17.72 [-42.77 to 7.34] | 8.16 [-18.72 to 35.04]
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = -20.00, 95% CI 2-sided [-52.73 to 12.74]
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = -24.70, 95% CI 2-sided [-50.80 to 1.39]
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = -22.61, 95% CI 2-sided [-53.39 to 8.16]
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = -31.67, 95% CI 2-sided [-63.44 to 0.09]
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = -5.79, 95% CI 2-sided [-38.33 to 26.74]

7. Secondary Outcome: Mean Change From Baseline at Week 16 in Serum Gamma Glutamyl Transferase (GGT), Among Those With a High Risk of PBC Progression
Description: as for outcome 5
Time Frame: Baseline and at Week 16
Population: High Risk Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: International Units per Liter
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 11 | 5 | 11 | 7 | 6 | 5
International Units per Liter | 47.5 [-9.9 to 104.8] | -58.5 [-142.5 to 25.5] | -18.0 [-74.9 to 38.9] | 4.6 [-66.5 to 75.8] | -18.4 [-93.6 to 56.8] | -6.7 [-89.1 to 75.8]
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = -106.0, 95% CI 2-sided [-205.1 to -6.8]
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = -65.5, 95% CI 2-sided [-148.5 to 17.6]
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = -42.8, 95% CI 2-sided [-136.5 to 50.9]
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = -65.8, 95% CI 2-sided [-161.2 to 29.5]
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = -54.1, 95% CI 2-sided [-153.6 to 45.3]

8. Secondary Outcome: Mean Change From Baseline at Week 16 in Total Bilirubin Concentration, Among Those With a High Risk of PBC Progression
Description: Baseline is the assessment performed at Week 4 (V3), or if missing then Visit 2 or Visit 1, excluding unscheduled visits. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Analysis was performed using ANCOVA including treatment group and Baseline.
Time Frame: Baseline and at Week 16
Population: High Risk Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Micromoles per Liter
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 11 | 5 | 11 | 7 | 6 | 5
Micromoles per Liter | 1.258 [-2.068 to 4.583] | -4.841 [-9.693 to 0.011] | -1.079 [-4.345 to 2.187] | -0.975 [-5.150 to 3.201] | -0.234 [-4.914 to 4.446] | 6.494 [1.622 to 11.365]
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = -6.099, 95% CI 2-sided [-11.929 to -0.268]
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = -2.337, 95% CI 2-sided [-6.962 to 2.289]
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = -2.232, 95% CI 2-sided [-7.679 to 3.215]
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = -1.492, 95% CI 2-sided [-7.413 to 4.430]
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = 5.236, 95% CI 2-sided [-0.591 to 11.063]

9. Secondary Outcome: Mean Change From Baseline at Week 16 in Albumin Concentration, Among Those With a High Risk of PBC Progression
Description: as for outcome 8
Time Frame: Baseline and at Week 16
Population: High Risk Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Grams per Liter
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 11 | 5 | 11 | 7 | 6 | 5
Grams per Liter | 0.0 [-1.2 to 1.3] | -0.5 [-2.3 to 1.3] | 0.3 [-1.0 to 1.6] | 0.8 [-0.8 to 2.3] | 0.0 [-1.7 to 1.7] | 0.7 [-1.1 to 2.5]
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = -0.5, 95% CI 2-sided [-2.7 to 1.6]
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = 0.3, 95% CI 2-sided [-1.5 to 2.1]
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = 0.7, 95% CI 2-sided [-1.2 to 2.7]
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = 0.0, 95% CI 2-sided [-2.1 to 2.0]
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = 0.7, 95% CI 2-sided [-1.5 to 2.9]

10. Secondary Outcome: Mean Change From Baseline at Week 16 in Prothrombin International Normalized Ratio (INR), Among Those With a High Risk of PBC Progression
Description: as for outcome 5
Time Frame: Baseline and at Week 16
Population: High Risk Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 9 | 5 | 11 | 6 | 7 | 5
Ratio | 0.01 [-0.03 to 0.05] | -0.01 [-0.06 to 0.04] | -0.03 [-0.06 to 0.00] | 0.01 [-0.04 to 0.05] | -0.02 [-0.07 to 0.02] | -0.03 [-0.08 to 0.02]
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = -0.02, 95% CI 2-sided [-0.08 to 0.04]
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.09 to 0.01]
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = 0.00, 95% CI 2-sided [-0.06 to 0.05]
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = -0.03, 95% CI 2-sided [-0.09 to 0.02]
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = -0.04, 95% CI 2-sided [-0.10 to 0.02]

11. Secondary Outcome: Mean Change From Baseline at Week 16 in Prothrombin Time, Among Those With a High Risk of PBC Progression
Description: as for outcome 5
Time Frame: Baseline and at Week 16
Population: High Risk Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Seconds
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 9 | 5 | 11 | 6 | 7 | 5
Seconds | -0.10 [-0.40 to 0.20] | 0.05 [-0.33 to 0.44] | -0.21 [-0.47 to 0.05] | 0.02 [-0.33 to 0.37] | -0.18 [-0.51 to 0.15] | -0.17 [-0.55 to 0.22]
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = 0.15, 95% CI 2-sided [-0.33 to 0.63]
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = -0.11, 95% CI 2-sided [-0.51 to 0.30]
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = 0.12, 95% CI 2-sided [-0.34 to 0.58]
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = -0.08, 95% CI 2-sided [-0.54 to 0.38]
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = -0.07, 95% CI 2-sided [-0.54 to 0.41]

12. Secondary Outcome: Number of Participants With Non-serious Adverse Events (Non-SAEs) and Serious Adverse Events (SAEs) -Main Study Period
Description: An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of a study treatment, whether or not considered related to the study treatment. Any untoward event resulting in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in persisting disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment is categorized as SAE.
Time Frame: Up to 12 weeks
Population: Safety Population. It consisted of all randomized participants who received at least 1 dose of study intervention.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo -Main Study Period: Eligible participants were randomized to receive GSK2330672 matching placebo via oral route for 12 weeks in Main Study Period.
- GSK2330672 20 mg QD - Main Study Period: Eligible participants were randomized to receive GSK2330672 20 milligrams (mg) once daily (QD) for 12 weeks in the Main Study period.
- GSK2330672 90 mg QD - Main Study Period: Eligible participants were randomized to receive GSK2330672 90 mg QD for 12 weeks in the Main study period.
- GSK2330672 180 mg QD - Main Study Period: Eligible participants were randomized to receive GSK2330672 180 mg QD for 12 weeks in the Main study period.
- GSK2330672 40 mg BID - Main Study Period: Eligible participants were randomized to receive GSK2330672 40 mg twice daily (BID) for 12 weeks in the Main study period.
- GSK2330672 90 mg BID - Main Study Period: Eligible participants were randomized to receive GSK2330672 90 mg BID for 12 weeks in the Main study period.
Arm/Group | Placebo -Main Study Period | GSK2330672 20 mg QD - Main Study Period | GSK2330672 90 mg QD - Main Study Period | GSK2330672 180 mg QD - Main Study Period | GSK2330672 40 mg BID - Main Study Period | GSK2330672 90 mg BID - Main Study Period
Number analyzed (Participants) | 36 | 16 | 23 | 27 | 23 | 22
Participants
  Any non-SAE | 17 | 11 | 19 | 24 | 16 | 18
  Any SAE | 0 | 0 | 1 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With Non-SAEs and SAEs -Final Study Period
Description: as for outcome 12
Time Frame: Up to 4 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Placebo - Final Study Period: Eligible participants were randomized to receive GSK2330672 matching placebo via oral route for 4 weeks in Final Study Period.
- GSK2330672 20 mg QD - Final Study Period: Eligible participants were randomized to receive GSK2330672 matching placebo via oral route for 4 weeks in Final Study Period. Participants received GSK2330672 20 mg QD during Main study period.
- GSK2330672 90 mg QD - Final Study Period: Eligible participants were randomized to receive GSK2330672 matching placebo via oral route for 4 weeks in Final Study Period. Participants received GSK2330672 90 mg QD during Main study period.
- GSK2330672 180 mg QD - Final Study Period: Eligible participants were randomized to receive GSK2330672 matching placebo via oral route for 4 weeks in Final Study Period. Participants received GSK2330672 180 mg QD during Main study period.
- GSK2330672 40 mg BID - Final Study Period: Eligible participants were randomized to receive GSK2330672 matching placebo via oral route for 4 weeks in Final Study Period. Participants received GSK2330672 40 mg BID during Main study period.
- GSK2330672 90 mg BID - Final Study Period: Eligible participants were randomized to receive GSK2330672 matching placebo via oral route for 4 weeks in Final Study Period. Participants received GSK2330672 90 mg BID during Main study period.
Arm/Group | Placebo - Final Study Period | GSK2330672 20 mg QD - Final Study Period | GSK2330672 90 mg QD - Final Study Period | GSK2330672 180 mg QD - Final Study Period | GSK2330672 40 mg BID - Final Study Period | GSK2330672 90 mg BID - Final Study Period
Number analyzed (Participants) | 35 | 16 | 19 | 19 | 21 | 17
Participants
  Any non-SAE | 2 | 6 | 8 | 2 | 2 | 2
  Any SAE | 0 | 0 | 0 | 0 | 0 | 0

14. Secondary Outcome: Number of Participants With Non-SAEs and SAEs - Follow-up Period
Description: as for outcome 12
Time Frame: Up to 4 weeks
Population: Safety Population
Measure: Count of Participants; unit: Participants
Groups:
- Placebo - Follow-up: Participants who received GSK2330672 matching placebo in Main study period and Final study period entered in a 4-week no-treatment follow-up period.
- GSK2330672 20 mg QD - Follow-up; GSK2330672 90 mg QD - Follow-up; GSK2330672 180 mg QD - Follow-up; GSK2330672 40 mg BID - Follow-up; GSK2330672 90 mg BID - Follow-up: Participants who received treatment (active or placebo) in Main study period and Final study period entered in a 4-week no-treatment follow-up period.
Arm/Group | Placebo - Follow-up | GSK2330672 20 mg QD - Follow-up | GSK2330672 90 mg QD - Follow-up | GSK2330672 180 mg QD - Follow-up | GSK2330672 40 mg BID - Follow-up | GSK2330672 90 mg BID - Follow-up
Number analyzed (Participants) | 35 | 16 | 23 | 27 | 22 | 22
Participants
  Any non-SAE | 0 | 0 | 0 | 0 | 0 | 0
  Any SAE | 0 | 1 | 0 | 1 | 0 | 0

15. Secondary Outcome: Number of Participants With Clinical Chemistry Data of Potential Clinical Importance
Description: Blood samples were collected to measure analyze the following parameters: albumin, calcium, Glomerular filtration rate (GFR) from creatinine, glucose, potassium and sodium. Participants were counted in the worst case category that their value changes to (low, within range [w/in] or no change, or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (for example [e.g.], high to high), or whose value became within range, were recorded in the "To w/in Range or No Change" category. Participants were counted twice if the participant had values that changed "To Low" and "To High", so the percentages may not add to 100 percent (%). Only "To Low" and/or "To High" categories with potential clinical importance data have been presented.
Time Frame: At Weeks 8, 12, 16 and 20
Population: Safety Population. Only those participants with data available at the specified data points were analyzed (represented by n= X in the category titles).
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 36 | 16 | 23 | 27 | 23 | 22
Participants
  Albumin, To Low, Week 8, n=36, 16, 21, 21, 22, 19: number analyzed (Participants) | 36 | 16 | 21 | 21 | 22 | 19
  Albumin, To Low, Week 8, n=36, 16, 21, 21, 22, 19 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin, To Low, Week 12, n=35, 16, 21, 23, 22, 21: number analyzed (Participants) | 35 | 16 | 21 | 23 | 22 | 21
  Albumin, To Low, Week 12, n=35, 16, 21, 23, 22, 21 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin, To Low, Week 16, n=35, 16, 21, 22, 21, 20: number analyzed (Participants) | 35 | 16 | 21 | 22 | 21 | 20
  Albumin, To Low, Week 16, n=35, 16, 21, 22, 21, 20 | 0 | 0 | 0 | 0 | 0 | 0
  Albumin, To Low, Week 20, n=35, 16, 22, 22, 22, 21: number analyzed (Participants) | 35 | 16 | 22 | 22 | 22 | 21
  Albumin, To Low, Week 20, n=35, 16, 22, 22, 22, 21 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium, To Low, Week 8, n=36, 16, 21, 21, 22, 19: number analyzed (Participants) | 36 | 16 | 21 | 21 | 22 | 19
  Calcium, To Low, Week 8, n=36, 16, 21, 21, 22, 19 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium, To High, Week 8, n=36, 16, 21, 21, 22, 19: number analyzed (Participants) | 36 | 16 | 21 | 21 | 22 | 19
  Calcium, To High, Week 8, n=36, 16, 21, 21, 22, 19 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium, To Low, Week 12, n=35, 16, 21, 23, 22, 21: number analyzed (Participants) | 35 | 16 | 21 | 23 | 22 | 21
  Calcium, To Low, Week 12, n=35, 16, 21, 23, 22, 21 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium, To High, Week 12, n=35, 16, 21, 23, 22, 21: number analyzed (Participants) | 35 | 16 | 21 | 23 | 22 | 21
  Calcium, To High, Week 12, n=35, 16, 21, 23, 22, 21 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium, To Low, Week 16, n=35, 16, 21, 22, 21, 20: number analyzed (Participants) | 35 | 16 | 21 | 22 | 21 | 20
  Calcium, To Low, Week 16, n=35, 16, 21, 22, 21, 20 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium, To High, Week 16, n=35, 16, 21, 22, 21, 20: number analyzed (Participants) | 35 | 16 | 21 | 22 | 21 | 20
  Calcium, To High, Week 16, n=35, 16, 21, 22, 21, 20 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium, To Low, Week 20, n=35, 16, 22, 22, 22, 21: number analyzed (Participants) | 35 | 16 | 22 | 22 | 22 | 21
  Calcium, To Low, Week 20, n=35, 16, 22, 22, 22, 21 | 0 | 0 | 0 | 0 | 0 | 0
  Calcium, To High, Week 20, n=35, 16, 22, 22, 22, 21: number analyzed (Participants) | 35 | 16 | 22 | 22 | 22 | 21
  Calcium, To High, Week 20, n=35, 16, 22, 22, 22, 21 | 1 | 0 | 0 | 0 | 0 | 0
  GFR, To Low, Week 8, n=36, 16, 21, 21, 22, 19: number analyzed (Participants) | 36 | 16 | 21 | 21 | 22 | 19
  GFR, To Low, Week 8, n=36, 16, 21, 21, 22, 19 | 0 | 0 | 0 | 0 | 0 | 0
  GFR, To Low, Week 12, n=35, 15, 21, 23, 22, 21: number analyzed (Participants) | 35 | 15 | 21 | 23 | 22 | 21
  GFR, To Low, Week 12, n=35, 15, 21, 23, 22, 21 | 0 | 0 | 0 | 0 | 0 | 0
  GFR, To Low, Week 16, n=35, 16, 21, 22, 21, 21: number analyzed (Participants) | 35 | 16 | 21 | 22 | 21 | 21
  GFR, To Low, Week 16, n=35, 16, 21, 22, 21, 21 | 0 | 0 | 0 | 0 | 0 | 0
  GFR, To Low, Week 20, n=35, 16, 22, 22, 22, 21: number analyzed (Participants) | 35 | 16 | 22 | 22 | 22 | 21
  GFR, To Low, Week 20, n=35, 16, 22, 22, 22, 21 | 0 | 0 | 0 | 1 | 0 | 0
  Glucose ,To Low, Week 8, n=36, 16, 21, 21, 22, 19: number analyzed (Participants) | 36 | 16 | 21 | 21 | 22 | 19
  Glucose ,To Low, Week 8, n=36, 16, 21, 21, 22, 19 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose ,To High, Week 8, n=36, 16, 21, 21, 22, 19: number analyzed (Participants) | 36 | 16 | 21 | 21 | 22 | 19
  Glucose ,To High, Week 8, n=36, 16, 21, 21, 22, 19 | 1 | 0 | 0 | 0 | 0 | 1
  Glucose ,To Low, Week 12, n=35, 16, 21, 23, 22, 21: number analyzed (Participants) | 35 | 16 | 21 | 23 | 22 | 21
  Glucose ,To Low, Week 12, n=35, 16, 21, 23, 22, 21 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose, To High, Week 12, n=35, 16, 21, 23, 22, 21: number analyzed (Participants) | 35 | 16 | 21 | 23 | 22 | 21
  Glucose, To High, Week 12, n=35, 16, 21, 23, 22, 21 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose ,To Low, Week 16, n=35, 16, 21, 22, 21,20: number analyzed (Participants) | 35 | 16 | 21 | 22 | 21 | 20
  Glucose ,To Low, Week 16, n=35, 16, 21, 22, 21,20 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose, To High, Week 16, n=35, 16, 21, 22, 21, 20: number analyzed (Participants) | 35 | 16 | 21 | 22 | 21 | 20
  Glucose, To High, Week 16, n=35, 16, 21, 22, 21, 20 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose ,To Low, Week 20, n=35, 16, 22, 22, 22, 21: number analyzed (Participants) | 35 | 16 | 22 | 22 | 22 | 21
  Glucose ,To Low, Week 20, n=35, 16, 22, 22, 22, 21 | 0 | 0 | 0 | 0 | 0 | 0
  Glucose, To High, Week 20, n=35, 16, 22, 22, 22, 21: number analyzed (Participants) | 35 | 16 | 22 | 22 | 22 | 21
  Glucose, To High, Week 20, n=35, 16, 22, 22, 22, 21 | 1 | 0 | 0 | 0 | 0 | 0
  Potassium,To Low, Week 8, n=36, 16, 21, 21, 22, 19: number analyzed (Participants) | 36 | 16 | 21 | 21 | 22 | 19
  Potassium,To Low, Week 8, n=36, 16, 21, 21, 22, 19 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium, To High, Week 8, n=36, 16, 21, 21, 22, 19: number analyzed (Participants) | 36 | 16 | 21 | 21 | 22 | 19
  Potassium, To High, Week 8, n=36, 16, 21, 21, 22, 19 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium,To Low, Week 12, n=35, 16, 21, 23, 22, 21: number analyzed (Participants) | 35 | 16 | 21 | 23 | 22 | 21
  Potassium,To Low, Week 12, n=35, 16, 21, 23, 22, 21 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium, To High, Week 12, n=35, 16, 21, 23, 22, 21: number analyzed (Participants) | 35 | 16 | 21 | 23 | 22 | 21
  Potassium, To High, Week 12, n=35, 16, 21, 23, 22, 21 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium,To Low, Week 16, n=35, 16, 21, 22, 21, 20: number analyzed (Participants) | 35 | 16 | 21 | 22 | 21 | 20
  Potassium,To Low, Week 16, n=35, 16, 21, 22, 21, 20 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium, To High, Week 16, n=35, 16, 21, 22, 21, 20: number analyzed (Participants) | 35 | 16 | 21 | 22 | 21 | 20
  Potassium, To High, Week 16, n=35, 16, 21, 22, 21, 20 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium,To Low, Week 20, n=35, 16, 22, 22, 22, 21: number analyzed (Participants) | 35 | 16 | 22 | 22 | 22 | 21
  Potassium,To Low, Week 20, n=35, 16, 22, 22, 22, 21 | 0 | 0 | 0 | 0 | 0 | 0
  Potassium, To High, Week 20, n=35, 16, 22,22, 22, 21: number analyzed (Participants) | 35 | 16 | 22 | 22 | 22 | 21
  Potassium, To High, Week 20, n=35, 16, 22,22, 22, 21 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium, To Low, Week 8, n=36, 16, 21, 21, 22, 19: number analyzed (Participants) | 36 | 16 | 21 | 21 | 22 | 19
  Sodium, To Low, Week 8, n=36, 16, 21, 21, 22, 19 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium, To High, Week 8, n=36, 16, 21, 21, 22, 19: number analyzed (Participants) | 36 | 16 | 21 | 21 | 22 | 19
  Sodium, To High, Week 8, n=36, 16, 21, 21, 22, 19 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium, To Low, Week 12, n=35, 16, 21, 23, 22, 21: number analyzed (Participants) | 35 | 16 | 21 | 23 | 22 | 21
  Sodium, To Low, Week 12, n=35, 16, 21, 23, 22, 21 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium, To High, Week 12, n=35, 16, 21, 23, 22, 21: number analyzed (Participants) | 35 | 16 | 21 | 23 | 22 | 21
  Sodium, To High, Week 12, n=35, 16, 21, 23, 22, 21 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium, To Low, Week 16, n=35, 16, 21, 22, 21, 20: number analyzed (Participants) | 35 | 16 | 21 | 22 | 21 | 20
  Sodium, To Low, Week 16, n=35, 16, 21, 22, 21, 20 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium, To High, Week 16, n=35, 16, 21, 22, 21, 20: number analyzed (Participants) | 35 | 16 | 21 | 22 | 21 | 20
  Sodium, To High, Week 16, n=35, 16, 21, 22, 21, 20 | 0 | 0 | 1 | 0 | 0 | 0
  Sodium, To Low, Week 20, n=35, 16, 22, 22, 22, 21: number analyzed (Participants) | 35 | 16 | 22 | 22 | 22 | 21
  Sodium, To Low, Week 20, n=35, 16, 22, 22, 22, 21 | 0 | 0 | 0 | 0 | 0 | 0
  Sodium, To High, Week 20, n=35, 16, 22, 22, 22, 21: number analyzed (Participants) | 35 | 16 | 22 | 22 | 22 | 21
  Sodium, To High, Week 20, n=35, 16, 22, 22, 22, 21 | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Number of Participants With Hematology Data of Potential Clinical Importance
Description: Blood samples were collected to analyze the following parameters: hematocrit, hemoglobin, leukocytes, lymphocytes, neutrophils and platelets. Participants were counted in the worst case category that their value changes to (low, w/in or no change, or high), unless there is no change in their category. Participants whose laboratory value category was unchanged (e.g., high to high), or whose value became within range, were recorded in the "To w/in Range or No Change" category. Participants were counted twice if the participant had values that changed "To Low" and "To High", so the percentages may not add to 100%. Only "To Low" and/or "To High" categories with potential clinical importance data have been presented.
Time Frame: At Weeks 8, 12, 16 and 20
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 36 | 16 | 23 | 27 | 23 | 22
Participants
  Hematocrit, To High, Week 8,n=36, 16, 21, 21, 22, 19: number analyzed (Participants) | 36 | 16 | 21 | 21 | 22 | 19
  Hematocrit, To High, Week 8,n=36, 16, 21, 21, 22, 19 | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit, To High, Week 12, n=33, 15, 21, 23, 22, 20: number analyzed (Participants) | 33 | 15 | 21 | 23 | 22 | 20
  Hematocrit, To High, Week 12, n=33, 15, 21, 23, 22, 20 | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit, To High, Week 16, n=35, 15, 21, 22, 21, 21: number analyzed (Participants) | 35 | 15 | 21 | 22 | 21 | 21
  Hematocrit, To High, Week 16, n=35, 15, 21, 22, 21, 21 | 0 | 0 | 0 | 0 | 0 | 0
  Hematocrit, To High, Week 20, n=34, 16, 22, 22, 22, 20: number analyzed (Participants) | 34 | 16 | 22 | 22 | 22 | 20
  Hematocrit, To High, Week 20, n=34, 16, 22, 22, 22, 20 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin, To High, Week 8,n=36,16, 21, 21, 22,19: number analyzed (Participants) | 36 | 16 | 21 | 21 | 22 | 19
  Hemoglobin, To High, Week 8,n=36,16, 21, 21, 22,19 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin, To High, Week 12, n=33,15, 21, 23, 22, 20: number analyzed (Participants) | 33 | 15 | 21 | 23 | 22 | 20
  Hemoglobin, To High, Week 12, n=33,15, 21, 23, 22, 20 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin, To High, Week 16, n=35, 15, 21, 22, 21, 21: number analyzed (Participants) | 35 | 15 | 21 | 22 | 21 | 21
  Hemoglobin, To High, Week 16, n=35, 15, 21, 22, 21, 21 | 0 | 0 | 0 | 0 | 0 | 0
  Hemoglobin, To High, Week 20, n=34,16, 22, 22, 22, 20: number analyzed (Participants) | 34 | 16 | 22 | 22 | 22 | 20
  Hemoglobin, To High, Week 20, n=34,16, 22, 22, 22, 20 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes, To Low, Week 8, n=36,15, 21, 21, 22,19: number analyzed (Participants) | 36 | 15 | 21 | 21 | 22 | 19
  Leukocytes, To Low, Week 8, n=36,15, 21, 21, 22,19 | 1 | 0 | 0 | 0 | 1 | 0
  Leukocytes,To High, Week 8, n=36,15, 21, 21, 22,19: number analyzed (Participants) | 36 | 15 | 21 | 21 | 22 | 19
  Leukocytes,To High, Week 8, n=36,15, 21, 21, 22,19 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes, To Low, Week 12, n=33,15, 21, 23, 22, 20: number analyzed (Participants) | 33 | 15 | 21 | 23 | 22 | 20
  Leukocytes, To Low, Week 12, n=33,15, 21, 23, 22, 20 | 1 | 1 | 1 | 0 | 0 | 0
  Leukocytes,To High, Week 12, n=33,15,21,23, 22, 20: number analyzed (Participants) | 33 | 15 | 21 | 23 | 22 | 20
  Leukocytes,To High, Week 12, n=33,15,21,23, 22, 20 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes, To Low, Week 16, n=34, 15, 21, 22, 20, 21: number analyzed (Participants) | 34 | 15 | 21 | 22 | 20 | 21
  Leukocytes, To Low, Week 16, n=34, 15, 21, 22, 20, 21 | 1 | 0 | 3 | 1 | 1 | 0
  Leukocytes,To High, Week 16, n=34, 15, 21, 22, 20, 21: number analyzed (Participants) | 34 | 15 | 21 | 22 | 20 | 21
  Leukocytes,To High, Week 16, n=34, 15, 21, 22, 20, 21 | 0 | 0 | 0 | 0 | 0 | 0
  Leukocytes, To Low, Week 20, n=34,16, 22, 21, 22, 19: number analyzed (Participants) | 34 | 16 | 22 | 21 | 22 | 19
  Leukocytes, To Low, Week 20, n=34,16, 22, 21, 22, 19 | 0 | 1 | 1 | 0 | 0 | 0
  Leukocytes, To High, Week 20, n=34,16, 22, 21, 22, 19: number analyzed (Participants) | 34 | 16 | 22 | 21 | 22 | 19
  Leukocytes, To High, Week 20, n=34,16, 22, 21, 22, 19 | 0 | 0 | 0 | 0 | 0 | 0
  Lymphocytes, To Low, Week 8, n=35,15, 21, 21, 22, 19: number analyzed (Participants) | 35 | 15 | 21 | 21 | 22 | 19
  Lymphocytes, To Low, Week 8, n=35,15, 21, 21, 22, 19 | 2 | 0 | 0 | 0 | 0 | 0
  Lymphocytes, To Low, Week 12, n=32,15,21,23, 22, 20: number analyzed (Participants) | 32 | 15 | 21 | 23 | 22 | 20
  Lymphocytes, To Low, Week 12, n=32,15,21,23, 22, 20 | 1 | 0 | 0 | 2 | 0 | 0
  Lymphocytes, To Low, Week 16, n=34, 15, 21, 22, 20, 21: number analyzed (Participants) | 34 | 15 | 21 | 22 | 20 | 21
  Lymphocytes, To Low, Week 16, n=34, 15, 21, 22, 20, 21 | 0 | 0 | 0 | 1 | 0 | 0
  Lymphocytes, To Low, Week 20, n=34,16, 22, 21, 22, 19: number analyzed (Participants) | 34 | 16 | 22 | 21 | 22 | 19
  Lymphocytes, To Low, Week 20, n=34,16, 22, 21, 22, 19 | 0 | 0 | 1 | 0 | 0 | 0
  Neutrophils, To Low, Week 8,n=35,15, 21, 21, 22, 19: number analyzed (Participants) | 35 | 15 | 21 | 21 | 22 | 19
  Neutrophils, To Low, Week 8,n=35,15, 21, 21, 22, 19 | 1 | 1 | 0 | 1 | 1 | 1
  Neutrophils, To Low, Week 12, n=32, 15, 21, 23, 22, 20: number analyzed (Participants) | 32 | 15 | 21 | 23 | 22 | 20
  Neutrophils, To Low, Week 12, n=32, 15, 21, 23, 22, 20 | 0 | 1 | 0 | 1 | 0 | 1
  Neutrophils, To Low, Week 16, n=34, 15, 21, 22, 20, 21: number analyzed (Participants) | 34 | 15 | 21 | 22 | 20 | 21
  Neutrophils, To Low, Week 16, n=34, 15, 21, 22, 20, 21 | 1 | 0 | 2 | 0 | 1 | 0
  Neutrophils, To Low, Week 20, n=34,16, 22, 21, 22,19: number analyzed (Participants) | 34 | 16 | 22 | 21 | 22 | 19
  Neutrophils, To Low, Week 20, n=34,16, 22, 21, 22,19 | 0 | 0 | 1 | 0 | 0 | 0
  Platelets, To Low, Week 8,n=36,15, 20, 21, 22,19: number analyzed (Participants) | 36 | 15 | 20 | 21 | 22 | 19
  Platelets, To Low, Week 8,n=36,15, 20, 21, 22,19 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets, To High, Week 8,n=36,15, 20, 21, 22, 19: number analyzed (Participants) | 36 | 15 | 20 | 21 | 22 | 19
  Platelets, To High, Week 8,n=36,15, 20, 21, 22, 19 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets, To Low, Week 12, n=33,14,19, 23, 22, 20: number analyzed (Participants) | 33 | 14 | 19 | 23 | 22 | 20
  Platelets, To Low, Week 12, n=33,14,19, 23, 22, 20 | 0 | 0 | 0 | 0 | 0 | 1
  Platelets,To High, Week 12, n=33, 14, 19, 23, 22, 20: number analyzed (Participants) | 33 | 14 | 19 | 23 | 22 | 20
  Platelets,To High, Week 12, n=33, 14, 19, 23, 22, 20 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets, To Low, Week 16, n=35, 14, 19, 22, 21, 21: number analyzed (Participants) | 35 | 14 | 19 | 22 | 21 | 21
  Platelets, To Low, Week 16, n=35, 14, 19, 22, 21, 21 | 1 | 0 | 0 | 0 | 0 | 1
  Platelets,To High, Week 16, n=35, 14, 19, 22, 21, 21: number analyzed (Participants) | 35 | 14 | 19 | 22 | 21 | 21
  Platelets,To High, Week 16, n=35, 14, 19, 22, 21, 21 | 1 | 0 | 0 | 0 | 0 | 0
  Platelets, To Low, Week 20, n=33,16, 21, 21, 22, 20: number analyzed (Participants) | 33 | 16 | 21 | 21 | 22 | 20
  Platelets, To Low, Week 20, n=33,16, 21, 21, 22, 20 | 0 | 0 | 0 | 0 | 0 | 0
  Platelets,To High, Week 20, n=33, 16, 21, 21, 22, 20: number analyzed (Participants) | 33 | 16 | 21 | 21 | 22 | 20
  Platelets,To High, Week 20, n=33, 16, 21, 21, 22, 20 | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Number of Participants With Abnormal 12-Lead Electrocardiogram (ECG) Parameters
Description: A 12-lead ECG was recorded with the participant in a semi-supine position. 12-lead ECGs were obtained by using an automated ECG machine. Data for abnormal, not clinically significant (NCS) and clinically significant (CS) ECG findings are presented. CS abnormal findings are those which are not associated with the underlying disease, unless judged by the investigator to be more severe than expected for the participant's condition.
Time Frame: At Weeks 8, 12, 16 and 20
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 36 | 16 | 23 | 27 | 23 | 22
Participants
  Abnormal, NCS, Week 8, n=36, 16, 21, 21, 22,19: number analyzed (Participants) | 36 | 16 | 21 | 21 | 22 | 19
  Abnormal, NCS, Week 8, n=36, 16, 21, 21, 22,19 | 10 | 2 | 1 | 7 | 8 | 4
  Abnormal, CS, Week 8, n=36, 16, 21, 21, 22, 19: number analyzed (Participants) | 36 | 16 | 21 | 21 | 22 | 19
  Abnormal, CS, Week 8, n=36, 16, 21, 21, 22, 19 | 0 | 0 | 0 | 1 | 0 | 0
  Abnormal, NCS, Week 12, n= 35, 16, 20, 23, 22, 21: number analyzed (Participants) | 35 | 16 | 20 | 23 | 22 | 21
  Abnormal, NCS, Week 12, n= 35, 16, 20, 23, 22, 21 | 9 | 3 | 3 | 8 | 8 | 4
  Abnormal, CS, Week 12, n=35, 16, 20, 23, 22, 21: number analyzed (Participants) | 35 | 16 | 20 | 23 | 22 | 21
  Abnormal, CS, Week 12, n=35, 16, 20, 23, 22, 21 | 0 | 0 | 0 | 0 | 0 | 0
  Abnormal, NCS, Week 16, n= 35, 16, 21, 21, 22 ,21: number analyzed (Participants) | 35 | 16 | 21 | 21 | 22 | 21
  Abnormal, NCS, Week 16, n= 35, 16, 21, 21, 22 ,21 | 9 | 3 | 2 | 5 | 7 | 4
  Abnormal, CS, Week 16, n=35, 16, 21, 21, 22, 21: number analyzed (Participants) | 35 | 16 | 21 | 21 | 22 | 21
  Abnormal, CS, Week 16, n=35, 16, 21, 21, 22, 21 | 0 | 0 | 0 | 0 | 0 | 0
  Abnormal, NCS, Week 20, n=35, 16, 22, 22, 22, 20: number analyzed (Participants) | 35 | 16 | 22 | 22 | 22 | 20
  Abnormal, NCS, Week 20, n=35, 16, 22, 22, 22, 20 | 8 | 3 | 2 | 7 | 8 | 3
  Abnormal, CS, Week 20, n=35, 16, 22, 22, 22, 20: number analyzed (Participants) | 35 | 16 | 22 | 22 | 22 | 20
  Abnormal, CS, Week 20, n=35, 16, 22, 22, 22, 20 | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: SBP and DBP were measured in the semi-supine position with a completely automated device after at least 5 minutes of rest for the participant in a quiet setting without distractions. Baseline is the assessment performed at Week 4 (V3), or if missing then Visit 2 or Visit 1, excluding unscheduled visits. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 20
Population: Safety Population. Only those participants with data available at the specified data points were analyzed .
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 35 | 16 | 22 | 22 | 22 | 21
Millimeters of mercury (mmHg)
  SBP | -3.3 (13.33) | -2.1 (11.47) | 0.1 (12.78) | 0.7 (10.42) | -0.3 (15.16) | 2.0 (15.43)
  DBP | -1.3 (8.99) | 0.3 (7.75) | -0.3 (9.16) | -0.7 (5.51) | 2.5 (8.64) | 2.3 (7.23)

19. Secondary Outcome: Change From Baseline in Pulse Rate
Description: Pulse rate was measured in a semi-supine position after 5 minutes of rest. Baseline is the assessment performed at Week 4 (V3), or if missing then Visit 2 or Visit 1, excluding unscheduled visits. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and Week 20
Population: Safety Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 35 | 16 | 22 | 22 | 22 | 21
Beats per minute | 1.5 (7.19) | -2.6 (10.35) | 1.2 (10.91) | -0.2 (7.93) | 3.4 (8.92) | 0.5 (8.03)

20. Secondary Outcome: Change From Baseline in Gastrointestinal Symptom Rating Scale (GSRS) Assessment
Description: GSRS is a validated scale used to assess gastrointestinal symptoms experienced by participants over the preceding 5 to 7 days. GSRS was measured for all 5 domains: Average Diarrhea Syndrome Score, Average Indigestion Syndrome Score, Average Constipation Syndrome Score, Average Abdominal Pain Syndrome Score, Average Reflux Syndrome Score. All individual domains are scored on a 7-point Likert scale ranging from 1(not at all) to 7(extremely). Higher score indicate more severe symptoms. The Average Total GSRS score was mean of these 5 domains and ranges from 1 to 7. Higher score indicates worst possible degree of symptoms. The responses summarized at each visit are those given during the week prior to the visit, with exception of Day 1. Baseline is the most recent assessment completed by participant prior to randomization. Change from Baseline was calculated as post-Baseline value minus the Baseline value. Data has been presented for each domain along with the average Total GSRS score.
Time Frame: Baseline and Week 20
Population: Safety Population. Only those participants with data available at the specified data points were analyzed .
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 33 | 16 | 20 | 21 | 22 | 20
Scores on a scale
  Average Diarrhea Syndrome Score | 0.22 (1.343) | 0.15 (1.587) | 0.23 (1.180) | -0.13 (0.637) | -0.23 (1.729) | 0.22 (1.565)
  Average Indigestion Syndrome Score | -0.01 (1.138) | 0.09 (0.865) | -0.03 (0.811) | -0.14 (0.820) | -0.31 (1.046) | -0.54 (1.007)
  Average Constipation Syndrome Score | -0.03 (1.045) | -0.15 (0.989) | 0.32 (1.370) | -0.02 (0.934) | -0.32 (1.215) | -0.37 (0.772)
  Average Abdominal Pain Syndrome Score | -0.05 (1.074) | 0.06 (0.712) | -0.02 (1.000) | -0.06 (0.629) | -0.08 (0.885) | -0.25 (0.904)
  Average Reflux Syndrome Score | -0.09 (1.208) | -0.13 (0.619) | -0.20 (1.332) | -0.26 (0.664) | -0.16 (0.762) | -0.43 (0.847)
  Average Total Score | 0.01 (0.830) | 0.02 (0.668) | 0.07 (0.802) | -0.11 (0.433) | -0.23 (0.690) | -0.28 (0.695)

21. Secondary Outcome: Number of Participants With Mean Worst Daily Itch Score of <4 at Week 16
Description: Participants were required to score the severity of their itching using a 0-10 NRS where 0 represents no itching and 10 indicates the worst imaginable itching. The Worst Daily Itch Score is the most severe (highest) NRS recorded on a given day. Mean Worst Daily Itch score was calculated as the average of the worst daily itch scores provided in the 7 days prior to the Week 16 visit. Number of participants with Mean Worst Daily Itch Score of <4 at Week 16 is presented.
Time Frame: At Week 16
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 36 | 16 | 23 | 27 | 23 | 22
Participants | 21 | 13 | 14 | 18 | 18 | 14
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Odds Ratio (OR) = 2.89, 95% CI 2-sided [0.69 to 12.02] — Analysis was performed using Logistic regression. No covariates were used
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Odds Ratio (OR) = 1.56, 95% CI 2-sided [0.48 to 5.02] — Analysis was performed using Logistic regression. No covariates were used
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Odds Ratio (OR) = 3.00, 95% CI 2-sided [0.84 to 10.76] — Analysis was performed using Logistic regression. No covariates were used
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Odds Ratio (OR) = 3.00, 95% CI 2-sided [0.84 to 10.76] — Analysis was performed using Logistic regression. No covariates were used
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Odds Ratio (OR) = 1.33, 95% CI 2-sided [0.43 to 4.13] — Analysis was performed using Logistic regression. No covariates were used

22. Secondary Outcome: Number of Participants With Improvement of >= 30 Percent (%) in the Mean Worst Daily Itch Score at Week 16 From Baseline
Description: Participants were required to score the severity of their itching using a 0-10 NRS where 0 represents no itching and 10 indicates the worst imaginable itching. The Worst Daily Itch Score is the most severe (highest) NRS recorded on a given day. Mean Worst Daily Itch score was calculated as the average of the worst daily itch scores provided in the 7 days prior to the Week 16 visit. Baseline is the most recent assessment completed by the participant prior to randomization. Number of participants with improvement of >= 30% in the Mean Worst Daily Itch Score at Week 16 from Baseline is presented.
Time Frame: Baseline and At Week 16
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 36 | 16 | 23 | 27 | 23 | 22
Participants | 17 | 9 | 15 | 14 | 15 | 14
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Odds Ratio (OR) = 1.36, 95% CI 2-sided [0.41 to 4.47] — Analysis was performed using Logistic regression. No covariates were used
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Odds Ratio (OR) = 3.18, 95% CI 2-sided [0.95 to 10.65] — Analysis was performed using Logistic regression. No covariates were used
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Odds Ratio (OR) = 1.85, 95% CI 2-sided [0.62 to 5.53] — Analysis was performed using Logistic regression. No covariates were used
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Odds Ratio (OR) = 2.27, 95% CI 2-sided [0.74 to 6.92] — Analysis was performed using Logistic regression. No covariates were used
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Odds Ratio (OR) = 2.12, 95% CI 2-sided [0.69 to 6.51] — Analysis was performed using Logistic regression. No covariates were used

23. Secondary Outcome: Number of Participants With Improvement of >=2 in the Mean Worst Daily Itch Score at Week 16 From Baseline
Description: Participants were required to score the severity of their itching using a 0-10 NRS where 0 represents no itching and 10 indicates the worst imaginable itching. The Worst Daily Itch Score is the most severe (highest) NRS recorded on a given day. Mean Worst Daily Itch score was calculated as the average of the worst daily itch scores provided in the 7 days prior to the Week 16 visit. Baseline is the most recent assessment completed by the participant prior to randomization. Number of participants with improvement of >=2 in the Mean Worst Daily Itch Score at Week 16 from Baseline is presented.
Time Frame: Baseline and At Week 16
Population: ITT Population
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 36 | 16 | 23 | 27 | 23 | 22
Participants | 14 | 6 | 12 | 9 | 13 | 12
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Odds Ratio (OR) = 0.90, 95% CI 2-sided [0.27 to 3.04] — Analysis was performed using Logistic regression. No covariates were used
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Odds Ratio (OR) = 2.25, 95% CI 2-sided [0.73 to 6.91] — Analysis was performed using Logistic regression. No covariates were used
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Odds Ratio (OR) = 1.04, 95% CI 2-sided [0.35 to 3.08] — Analysis was performed using Logistic regression. No covariates were used
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Odds Ratio (OR) = 2.17, 95% CI 2-sided [0.73 to 6.42] — Analysis was performed using Logistic regression. No covariates were used
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Odds Ratio (OR) = 2.00, 95% CI 2-sided [0.67 to 5.99] — Analysis was performed using Logistic regression. No covariates were used

24. Secondary Outcome: Percentage of Responder Days With Worst Daily Itch Score of <4
Description: Percentage of Responder Days with Worst Daily Itch score was calculated as: (number of days response from Visit 3+1 to Visit 6-1 divided by number of days from Visit 3+1 to Visit 6-1 with worst daily itch scores available) times 100. Days for which no worst daily itch score was available did not contribute to either the numerator or the denominator. Analysis was performed using ANCOVA model including treatment group. Percentage of responder days with Worst Daily Itch Score of <4 is presented.
Time Frame: Up to Week 16
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of days
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 36 | 16 | 23 | 27 | 23 | 22
Percentage of days | 40.32 [28.79 to 51.86] | 58.53 [41.23 to 75.83] | 51.38 [36.95 to 65.81] | 58.76 [45.45 to 72.08] | 65.80 [51.37 to 80.23] | 53.58 [38.83 to 68.34]
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = 18.21, 95% CI 2-sided [-2.59 to 39.00]
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = 11.05, 95% CI 2-sided [-7.42 to 29.53]
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = 18.44, 95% CI 2-sided [0.82 to 36.06]
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = 25.48, 95% CI 2-sided [7.00 to 43.95]
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = 13.26, 95% CI 2-sided [-5.47 to 31.99]

25. Secondary Outcome: Percentage of Responder Days With Improvement of >= 30% in the Mean Worst Daily Itch Score at Week 16 From Baseline
Description: Percentage of Responder Days with Worst Daily Itch score was calculated as: (number of days response from Visit 3+1 to Visit 6-1 divided by number of days from Visit 3+1 to Visit 6-1 with worst daily itch scores available) times 100. Days for which no worst daily itch score was available did not contribute to either the numerator or the denominator. Analysis was performed using ANCOVA model including treatment group. Baseline is the most recent assessment completed by the participant prior to randomization. Percentage of responder days with improvement of >= 30% in the Mean Worst Daily Itch Score at Week 16 from Baseline is presented..
Time Frame: Baseline and at Week 16
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of days
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 36 | 16 | 23 | 27 | 23 | 22
Percentage of days | 38.46 [27.30 to 49.61] | 53.44 [36.71 to 70.18] | 45.43 [31.47 to 59.39] | 50.23 [37.35 to 63.12] | 60.29 [46.33 to 74.25] | 60.03 [45.76 to 74.31]
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = 14.99, 95% CI 2-sided [-5.13 to 35.10]
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = 6.97, 95% CI 2-sided [-10.90 to 24.84]
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = 11.78, 95% CI 2-sided [-5.27 to 28.82]
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = 21.83, 95% CI 2-sided [3.96 to 39.70]
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = 21.58, 95% CI 2-sided [3.46 to 39.69]

26. Secondary Outcome: Percentage of Responder Days With Improvement of >=2 in the Mean Worst Daily Itch Score at Week 16 From Baseline
Description: Percentage of Responder Days with Worst Daily Itch was calculated as: (number of days response from Visit 3+1 to Visit 6-1 divided by number of days from Visit 3+1 to Visit 6-1 with worst daily itch scores available) times 100. Days for which no worst daily itch score was available did not contribute to either the numerator or the denominator. Analysis was performed using ANCOVA model including treatment group. Baseline is the most recent assessment completed by the participant prior to randomization. Percentage of responder days with improvement of >=2 in the Mean Worst Daily Itch Score at Week 16 from Baseline is presented.
Time Frame: Baseline and at Week 16
Population: ITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of days
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 36 | 16 | 23 | 27 | 23 | 22
Percentage of days | 31.56 [19.96 to 43.16] | 37.71 [20.31 to 55.11] | 38.82 [24.31 to 53.33] | 40.69 [27.29 to 54.08] | 51.49 [36.98 to 66.00] | 58.60 [43.76 to 73.43]
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = 6.15, 95% CI 2-sided [-14.76 to 27.06]
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = 7.26, 95% CI 2-sided [-11.32 to 25.84]
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = 9.13, 95% CI 2-sided [-8.59 to 26.85]
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = 19.94, 95% CI 2-sided [1.36 to 38.51]
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = 27.04, 95% CI 2-sided [8.20 to 45.87]

27. Secondary Outcome: Change From Baseline in the Mean Daily Sleep Score at Week 16
Description: Mean Daily Sleep Score is defined as the average of the daily sleep scores provided in the 7 days prior to the relevant visit. Participants sleep quality was recorded in an electronic diary each morning using a 0-10 NRS in which 0: good sleep to 10:worst possible sleep. Higher score indicates worse possible sleep. Baseline is the average of the scores in the 7 days prior to the Week 4 (V3) visit. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Analysis was performed using ANCOVA including treatment group and Baseline.
Time Frame: Baseline and at Week 16
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 35 | 16 | 20 | 22 | 22 | 20
Scores on a scale | -1.39 [-2.06 to -0.72] | -1.66 [-2.64 to -0.67] | -1.87 [-2.75 to -0.99] | -1.85 [-2.69 to -1.01] | -2.35 [-3.19 to -1.50] | -1.69 [-2.57 to -0.81]
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = -0.27, 95% CI 2-sided [-1.46 to 0.92]
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = -0.48, 95% CI 2-sided [-1.58 to 0.62]
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = -0.46, 95% CI 2-sided [-1.53 to 0.61]
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = -0.96, 95% CI 2-sided [-2.03 to 0.12]
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = -0.30, 95% CI 2-sided [-1.40 to 0.80]

28. Secondary Outcome: Change From Baseline in the Mean Daily Fatigue Score at Week 16
Description: Mean Daily Fatigue Score is defined as the average of the daily fatigue scores provided in the 7 days prior to the relevant visit. Participants fatigue level was recorded in an electronic diary each evening using a 0-10 NRS in which 0: no fatigue to 10:worst possible fatigue. Higher score indicates worse possible fatigue. Baseline is the average of the scores in the 7 days prior to the Week 4 (V3) visit. Change from Baseline was calculated as the post-Baseline value minus the Baseline value. Analysis was performed using ANCOVA model including treatment group and Baseline.
Time Frame: Baseline and at Week 16
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 35 | 16 | 20 | 22 | 22 | 21
Scores on a scale | -0.79 [-1.39 to -0.18] | -1.18 [-2.08 to -0.27] | -1.19 [-2.00 to -0.37] | -1.04 [-1.81 to -0.28] | -1.20 [-1.97 to -0.44] | -1.07 [-1.86 to -0.29]
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = -0.39, 95% CI 2-sided [-1.49 to 0.71]
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = -0.40, 95% CI 2-sided [-1.41 to 0.61]
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = -0.26, 95% CI 2-sided [-1.24 to 0.72]
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = -0.42, 95% CI 2-sided [-1.39 to 0.56]
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = -0.29, 95% CI 2-sided [-1.28 to 0.70]

29. Secondary Outcome: Change From Baseline in the Five-Dimensional (5-D) Itch Scale at Week 16
Description: The 5-D itch scale had been developed as a brief, single page, instrument for the multidimensional quantification of itch that is sensitive to change over time. It has data to support its validity in a population of participants with pruritus and covers five dimensions of itch experienced by participants: duration, degree, direction, disability and distribution. Each domain was scored on a 5-point scale, ranging from 1 (Not present/resolved/never) to 5 (unbearable/getting worse/always), higher scores indicates worst itching. The scores of each of five domains were achieved separately and then summed together to obtain a total 5-D score. A total 5-D scores potentially ranged between 5 (no pruritus) and 25 (most severe pruritus) where higher score indicates worse possible itching. Baseline is assessment performed at Week 4 (V3) which is conducted prior to first dosing of randomized medication that evening. Change from Baseline was calculated as post-Baseline value minus Baseline value.
Time Frame: Baseline and at Week 16
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 35 | 16 | 21 | 21 | 22 | 20
Scores on a scale
  Duration | -0.8 [-1.1 to -0.4] | -0.9 [-1.3 to -0.4] | -0.4 [-0.8 to 0.0] | -1.2 [-1.6 to -0.8] | -0.6 [-1.0 to -0.2] | -0.7 [-1.1 to -0.3]
  Degree | -0.7 [-1.0 to -0.4] | -0.9 [-1.4 to -0.5] | -0.7 [-1.1 to -0.3] | -0.7 [-1.2 to -0.3] | -0.9 [-1.3 to -0.5] | -0.8 [-1.2 to -0.4]
  Direction | -0.7 [-1.1 to -0.3] | -0.7 [-1.3 to -0.1] | -0.7 [-1.2 to -0.2] | -0.9 [-1.4 to -0.4] | -1.1 [-1.6 to -0.6] | -0.7 [-1.2 to -0.2]
  Disability | -0.4 [-0.7 to 0.0] | -0.8 [-1.4 to -0.2] | -0.5 [-1.0 to 0.0] | -0.7 [-1.2 to -0.2] | -0.7 [-1.2 to -0.2] | -0.7 [-1.2 to -0.1]
  Distribution | -0.4 [-0.7 to -0.1] | -0.7 [-1.2 to -0.2] | -0.7 [-1.1 to -0.3] | -0.9 [-1.3 to -0.5] | -0.7 [-1.2 to -0.3] | -0.6 [-1.0 to -0.2]
  5-D Itch Total Score | -3.0 [-4.2 to -1.7] | -4.0 [-5.9 to -2.0] | -3.0 [-4.7 to -1.3] | -4.4 [-6.0 to -2.7] | -3.8 [-5.4 to -2.2] | -3.5 [-5.2 to -1.8]
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.7 to 0.5] — Duration
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = 0.4, 95% CI 2-sided [-0.2 to 0.9] — Duration
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = -0.4, 95% CI 2-sided [-1.0 to 0.1] — Duration
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = 0.2, 95% CI 2-sided [-0.3 to 0.7] — Duration
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = 0.1, 95% CI 2-sided [-0.4 to 0.6] — Duration
Statistical Analysis 6: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.8 to 0.3] — Degree
Statistical Analysis 7: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.5 to 0.5] — Degree
Statistical Analysis 8: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = -0.1, 95% CI 2-sided [-0.6 to 0.5] — Degree
Statistical Analysis 9: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.7 to 0.3] — Degree
Statistical Analysis 10: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Median Difference (Net) = -0.1, 95% CI 2-sided [-0.6 to 0.4] — Degree
Statistical Analysis 11: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.7 to 0.7] — Direction
Statistical Analysis 12: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.7 to 0.6] — Direction
Statistical Analysis 13: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.8 to 0.5] — Direction
Statistical Analysis 14: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = -0.4, 95% CI 2-sided [-1.0 to 0.2] — Direction
Statistical Analysis 15: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = 0.0, 95% CI 2-sided [-0.6 to 0.6] — Direction
Statistical Analysis 16: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = -0.4, 95% CI 2-sided [-1.1 to 0.3] — Disability
Statistical Analysis 17: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.8 to 0.5] — Disability
Statistical Analysis 18: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = -0.3, 95% CI 2-sided [-1.0 to 0.3] — Disability
Statistical Analysis 19: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = -0.3, 95% CI 2-sided [-1.0 to 0.3] — Disability
Statistical Analysis 20: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = -0.3, 95% CI 2-sided [-1.0 to 0.3] — Disability
Statistical Analysis 21: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.9 to 0.3] — Distribution
Statistical Analysis 22: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Median Difference (Net) = -0.3, 95% CI 2-sided [-0.9 to 0.2] — Distribution
Statistical Analysis 23: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = -0.5, 95% CI 2-sided [-1.0 to 0.0] — Distribution
Statistical Analysis 24: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = -0.3, 95% CI 2-sided [-0.9 to 0.2] — Distribution
Statistical Analysis 25: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = -0.2, 95% CI 2-sided [-0.7 to 0.3] — Distribution
Statistical Analysis 26: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = -1.0, 95% CI 2-sided [-3.3 to 1.3] — 5-D Itch Total Score
Statistical Analysis 27: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = -0.1, 95% CI 2-sided [-2.2 to 2.1] — 5-D Itch Total Score
Statistical Analysis 28: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = -1.4, 95% CI 2-sided [-3.5 to 0.7] — 5-D Itch Total Score
Statistical Analysis 29: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = -0.9, 95% CI 2-sided [-3.0 to 1.2] — 5-D Itch Total Score
Statistical Analysis 30: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = -0.6, 95% CI 2-sided [-2.7 to 1.6] — 5-D Itch Total Score

30. Secondary Outcome: Mean Change From Baseline at Week 16 in Serum Total Bile Acid Concentration
Description: Blood samples were collected for evaluating total bile acid concentration as a biomarker of PBC. Baseline is the assessment performed at Week 4 (V3), or if missing then Visit 2 or Visit 1, excluding unscheduled visits. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and at Week 16
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per Liter
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 35 | 16 | 20 | 22 | 21 | 21
Micromoles per Liter | -4.274 (20.0163) | -0.469 (6.5466) | -3.878 (40.1857) | -1.114 (6.9359) | -2.133 (8.9308) | 7.379 (38.8282)

31. Secondary Outcome: Mean Change From Baseline at Week 16 in Serum 7-alpha Hydroxy-4-cholesten-3-one (C4)
Description: Blood samples were collected for evaluating C4 concentration as a marker of bile acid synthesis. Baseline is the assessment performed at Week 4 (V3), or if missing then Visit 2 or Visit 1, excluding unscheduled visits. Change from Baseline was calculated as the post-Baseline value minus the Baseline value.
Time Frame: Baseline and at Week 16
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Micrograms per Liter
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 35 | 15 | 21 | 22 | 22 | 20
Micrograms per Liter | 4.746 (11.5644) | 10.703 (24.6045) | 11.452 (16.6371) | 29.488 (38.7584) | 58.674 (59.4833) | 40.629 (36.2769)

32. Secondary Outcome: Plasma Concentration of GSK2330672 After Sparse Sampling
Description: Blood samples were collected for measurement of plasma GSK2330672 concentration.
Time Frame: At Week 4 (between 1 and 3 hours post-dose) and At Weeks 8, 12 and 16 (between 1 and 3 hours post-dose, and between 5 and 8 hours post-dose)
Population: Pharmacokinetic (PK) Population consisted of any randomized participant who had at least one PK sample. Only those participants with data available at the specified data points were analyzed (represented by n=X in category titles).
Measure: Mean (Standard Deviation); unit: Picograms per milliliter
Arm/Group | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 16 | 23 | 27 | 23 | 22
Picograms per milliliter
  Week 4, Between 1 and 3 hours post-dose, n=6, 2, 7, 0, 4: number analyzed (Participants) | 6 | 2 | 7 | 0 | 4
  Week 4, Between 1 and 3 hours post-dose, n=6, 2, 7, 0, 4 | 5.00 (NA) — Standard deviation could not be calculated as >30% of samples were below the limit of quantification | 5.00 (NA) — Standard deviation could not be calculated as >30% of samples were below the limit of quantification | 32.71 (73.325) |  | 5.00 (NA) — Standard deviation could not be calculated as >30% of samples were below the limit of quantification
  Week 8, Between 1 and 3 hours post-dose, n=16, 21, 20, 22, 17: number analyzed (Participants) | 16 | 21 | 20 | 22 | 17
  Week 8, Between 1 and 3 hours post-dose, n=16, 21, 20, 22, 17 | 358.04 (665.685) | 958.81 (1563.265) | 2327.58 (3737.965) | 453.45 (967.424) | 2908.06 (5106.895)
  Week 8, Between 5 and 8 hours post-dose, n=14, 17, 18, 21, 16: number analyzed (Participants) | 14 | 17 | 18 | 21 | 16
  Week 8, Between 5 and 8 hours post-dose, n=14, 17, 18, 21, 16 | 300.04 (356.268) | 820.87 (1143.023) | 2234.28 (3420.442) | 339.74 (357.914) | 1990.89 (4061.978)
  Week 12, Between 1 and 3 hours post-dose, n=14, 19, 17, 20, 14: number analyzed (Participants) | 14 | 19 | 17 | 20 | 14
  Week 12, Between 1 and 3 hours post-dose, n=14, 19, 17, 20, 14 | 447.88 (1160.518) | 1594.16 (3133.370) | 2060.51 (2888.033) | 419.47 (774.321) | 3531.36 (6296.828)
  Week 12, Between 5 and 8 hours post-dose, n=14, 16, 17, 20, 13: number analyzed (Participants) | 14 | 16 | 17 | 20 | 13
  Week 12, Between 5 and 8 hours post-dose, n=14, 16, 17, 20, 13 | 341.39 (638.359) | 1084.00 (1353.089) | 2569.00 (3727.883) | 303.83 (300.716) | 2197.16 (3604.704)
  Week 16, Between 1 and 3 hours post-dose, n=3, 5, 4, 2, 5: number analyzed (Participants) | 3 | 5 | 4 | 2 | 5
  Week 16, Between 1 and 3 hours post-dose, n=3, 5, 4, 2, 5 | 394.00 (162.151) | 864.26 (1045.467) | 3328.50 (3185.646) | 338.50 (236.881) | 703.60 (756.010)
  Week 16, Between 5 and 8 hours post-dose, n=3, 3, 4, 2, 5: number analyzed (Participants) | 3 | 3 | 4 | 2 | 5
  Week 16, Between 5 and 8 hours post-dose, n=3, 3, 4, 2, 5 | 296.33 (118.154) | 578.00 (651.263) | 1940.50 (1128.203) | 364.50 (217.082) | 869.40 (1148.331)

33. Post Hoc Outcome: Mean Change From Baseline in Monthly Itch Score
Description: Participants were required to score severity of their itching each morning and evening using a 0-10 NRS where 0(no itching) and 10(worst imaginable itching). The worst of these 2 scores was Worst Daily Itch Score. For each week, mean Worst Daily Itch Score was calculated to form Mean Worst Daily Itch Score. The Monthly Itch Score was defined as worst weekly score (e.g., Mean Worst Daily Itch Score) for that month. The monthly itch score ranges from 0 to 10, higher score indicates worst imaginable itching. Baseline is average of scores in the 7 days prior to Week 4 (Visit 3 [V3]). Change from Baseline was calculated as post-Baseline value minus Baseline value. Mean change from Baseline in monthly itch score over 12 week treatment period is presented. Analysis was performed on change in Monthly Itch Scores over 12 week treatment period using Mixed model repeated measures (MMRM) with Baseline itch, treatment group, visit and a treatment group*visit interaction as covariates in the model.
Time Frame: Baseline and up to Week 12
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 36 | 16 | 23 | 24 | 22 | 22
Scores on a scale | -0.46 [-1.01 to 0.08] | -1.17 [-1.99 to -0.35] | -1.08 [-1.77 to -0.39] | -1.36 [-2.03 to -0.69] | -1.63 [-2.32 to -0.93] | -1.41 [-2.13 to -0.7]
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Mean Difference (Net) = -0.71, 95% CI 2-sided [-1.69 to 0.28]
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; Mean Difference (Net) = -0.62, 95% CI 2-sided [-1.49 to 0.26]
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; Mean Difference (Net) = -0.9, 95% CI 2-sided [-1.76 to -0.03]
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; Mean Difference (Net) = -1.16, 95% CI 2-sided [-2.05 to -0.28]
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; Mean Difference (Net) = -0.95, 95% CI 2-sided [-1.85 to -0.06]

34. Post Hoc Outcome: Ratio to Baseline in Total Serum Bile Acid Concentration
Description: Blood samples were collected for evaluation of total bile acid concentration as a biomarker of PBC. Baseline is the assessment performed at Week 4 (V3), or if missing then Visit 2 (Day 1) or Visit 1 (Screening), excluding unscheduled visits. Ratio to Baseline was defined as the geometric mean of post-Baseline visit value divided by the geometric mean of Baseline value. Values were log-transformed and mean change from Baseline on the log-scale was calculated over the 12 week treatment period. Analysis was performed on change in total serum bile acid concentration on the log-scale over the 12 week treatment period using Mixed model repeated measures (MMRM) with log-transformed Baseline total serum bile acid, visit, treatment group, a log-transformed Baseline total serum bile acid*visit interaction, and a treatment group*visit interaction used as covariates in the model. Afterwards, values were back-transformed to the original scale. Ratios of geometric means are presented.
Time Frame: Baseline and up to Week 12
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 36 | 16 | 22 | 24 | 22 | 22
Ratio | 1.01 [0.801 to 1.273] | 0.977 [0.688 to 1.386] | 1.182 [0.874 to 1.6] | 0.918 [0.687 to 1.226] | 0.697 [0.519 to 0.938] | 0.833 [0.616 to 1.127]
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; Least Square (LS) mean ratio = 0.967, 95% CI 2-sided [0.635 to 1.471]
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; LS mean ratio = 1.17, 95% CI 2-sided [0.8 to 1.712]
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; LS mean ratio = 0.909, 95% CI 2-sided [0.627 to 1.316]
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; LS mean ratio = 0.69, 95% CI 2-sided [0.474 to 1.005]
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; LS mean ratio = 0.825, 95% CI 2-sided [0.564 to 1.207]

35. Post Hoc Outcome: Ratio to Baseline in Serum 7-alpha-hydroxy-4-cholesten-3-one (C4) Concentration
Description: Blood samples were collected for evaluation of C4 concentration as a marker of bile acid synthesis. Baseline is the assessment performed at Week 4 (V3), or if missing then Visit 2 (Day 1) or Visit 1 (Screening), excluding unscheduled visits. Ratio to Baseline was defined as the geometric mean of post-Baseline visit value divided by the geometric mean of Baseline value. Values were log-transformed and mean change from Baseline on the log-scale was calculated over the 12 week treatment period. Analysis was performed on change in C4 on the log-scale over the 12 week treatment period using Mixed model repeated measures (MMRM) with log-transformed Baseline C4, visit, treatment group, a log-transformed Baseline C4*visit interaction, and a treatment group*visit interaction used as covariates in the model. Afterwards, values were back-transformed to the original scale. Ratios of geometric means are presented.
Time Frame: Baseline and up to Week 12
Population: ITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Least Squares Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Placebo | GSK2330672 20 mg QD | GSK2330672 90 mg QD | GSK2330672 180 mg QD | GSK2330672 40 mg BID | GSK2330672 90 mg BID
Number analyzed (Participants) | 36 | 16 | 22 | 24 | 22 | 22
Ratio | 1.158 [0.937 to 1.431] | 1.579 [1.151 to 2.166] | 2.374 [1.812 to 3.109] | 2.846 [2.192 to 3.694] | 3.622 [2.753 to 4.764] | 3.127 [2.385 to 4.101]
Statistical Analysis 1: Comparison: Placebo vs GSK2330672 20 mg QD; Test type: Other; LS mean ratio = 1.363, 95% CI 2-sided [0.932 to 1.995]
Statistical Analysis 2: Comparison: Placebo vs GSK2330672 90 mg QD; Test type: Other; LS mean ratio = 2.05, 95% CI 2-sided [1.456 to 2.887]
Statistical Analysis 3: Comparison: Placebo vs GSK2330672 180 mg QD; Test type: Other; LS mean ratio = 2.457, 95% CI 2-sided [1.758 to 3.436]
Statistical Analysis 4: Comparison: Placebo vs GSK2330672 40 mg BID; Test type: Other; LS mean ratio = 3.128, 95% CI 2-sided [2.206 to 4.435]
Statistical Analysis 5: Comparison: Placebo vs GSK2330672 90 mg BID; Test type: Other; LS mean ratio = 2.701, 95% CI 2-sided [1.915 to 3.81]

ADVERSE EVENTS:
Time Frame: Non-serious adverse events (Non-SAEs) and serious adverse events (SAEs) were collected up to 12 weeks during Main study period; up to 4 weeks during Final study period and up to 4 weeks during Follow-up period.
Description: Safety Population consisted of all randomized participants who received at least 1 dose of study intervention.
Groups:
- Placebo - Main Study Period: Eligible participants were randomized to receive GSK2330672 matching placebo via oral route for 12 weeks in Main Study Period.
Arm/Group | Placebo - Main Study Period | GSK2330672 20 mg QD - Main Study Period | GSK2330672 90 mg QD - Main Study Period | GSK2330672 180 mg QD - Main Study Period | GSK2330672 40 mg BID - Main Study Period | GSK2330672 90 mg BID - Main Study Period | Placebo - Final Study Period | GSK2330672 20 mg QD - Final Study Period | GSK2330672 90 mg QD - Final Study Period | GSK2330672 180 mg QD - Final Study Period | GSK2330672 40 mg BID - Final Study Period | GSK2330672 90 mg BID - Final Study Period | Placebo - Follow-up | GSK2330672 20 mg QD - Follow-up | GSK2330672 90 mg QD - Follow-up | GSK2330672 180 mg QD - Follow-up | GSK2330672 40 mg BID - Follow-up | GSK2330672 90 mg BID - Follow-up
All-Cause Mortality (participants affected / at risk) | 0/36 | 0/16 | 0/23 | 0/27 | 0/23 | 0/22 | 0/35 | 0/16 | 0/19 | 0/19 | 0/21 | 0/17 | 0/35 | 0/16 | 0/23 | 0/27 | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/16 | 1/23 | 0/27 | 0/23 | 0/22 | 0/35 | 0/16 | 0/19 | 0/19 | 0/21 | 0/17 | 0/35 | 1/16 | 0/23 | 1/27 | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 17/36 | 11/16 | 19/23 | 24/27 | 16/23 | 18/22 | 2/35 | 6/16 | 8/19 | 2/19 | 2/21 | 2/17 | 0/35 | 0/16 | 0/23 | 0/27 | 0/22 | 0/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Main Study Period (N=36) | GSK2330672 20 mg QD - Main Study Period (N=16) | GSK2330672 90 mg QD - Main Study Period (N=23) | GSK2330672 180 mg QD - Main Study Period (N=27) | GSK2330672 40 mg BID - Main Study Period (N=23) | GSK2330672 90 mg BID - Main Study Period (N=22) | Placebo - Final Study Period (N=35) | GSK2330672 20 mg QD - Final Study Period (N=16) | GSK2330672 90 mg QD - Final Study Period (N=19) | GSK2330672 180 mg QD - Final Study Period (N=19) | GSK2330672 40 mg BID - Final Study Period (N=21) | GSK2330672 90 mg BID - Final Study Period (N=17) | Placebo - Follow-up (N=35) | GSK2330672 20 mg QD - Follow-up (N=16) | GSK2330672 90 mg QD - Follow-up (N=23) | GSK2330672 180 mg QD - Follow-up (N=27) | GSK2330672 40 mg BID - Follow-up (N=22) | GSK2330672 90 mg BID - Follow-up (N=22)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo - Main Study Period (N=36) | GSK2330672 20 mg QD - Main Study Period (N=16) | GSK2330672 90 mg QD - Main Study Period (N=23) | GSK2330672 180 mg QD - Main Study Period (N=27) | GSK2330672 40 mg BID - Main Study Period (N=23) | GSK2330672 90 mg BID - Main Study Period (N=22) | Placebo - Final Study Period (N=35) | GSK2330672 20 mg QD - Final Study Period (N=16) | GSK2330672 90 mg QD - Final Study Period (N=19) | GSK2330672 180 mg QD - Final Study Period (N=19) | GSK2330672 40 mg BID - Final Study Period (N=21) | GSK2330672 90 mg BID - Final Study Period (N=17) | Placebo - Follow-up (N=35) | GSK2330672 20 mg QD - Follow-up (N=16) | GSK2330672 90 mg QD - Follow-up (N=23) | GSK2330672 180 mg QD - Follow-up (N=27) | GSK2330672 40 mg BID - Follow-up (N=22) | GSK2330672 90 mg BID - Follow-up (N=22)
Abdominal pain (Gastrointestinal disorders) | 3 (3) | 3 (3) | 4 (6) | 8 (9) | 2 (2) | 4 (5) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 2 (4) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asthenia (General disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone fissure (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 4 (5) | 6 (8) | 15 (20) | 18 (22) | 12 (14) | 15 (15) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 3 (3) | 1 (1) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingivitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 3 (5) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Impaired healing (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infectious mononucleosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 1 (2) | 1 (1) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin bacterial infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sleep disorder (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vitamin A deficiency (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-12-06): https://cdn.clinicaltrials.gov/large-docs/34/NCT02966834/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-14): https://cdn.clinicaltrials.gov/large-docs/34/NCT02966834/SAP_001.pdf